CLINICAL TRIAL: NCT00826007
Title: Associated Factors in Perioperative Hypoglycemia in Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Collaborators: Oakland University (Other)
Responsible Party: Principal Investigator, Tamra Dukatz, CRNA, Anesthesia Department, Corewell Health East
Other Study IDs: 2008-281
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes; Hypoglycemia
Keywords: perioperative hypoglycemia diabetes surgery; surgery
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: None Retained — non applicable
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to review incidences of mild, moderate, and severe hypoglycemia in preoperative care units, operating rooms, and postanesthesia care units and analyze associated conditions and treatment.

DETAILED DESCRIPTION:
With evidence linking surgical morbidity to hyperglycemia (high blood sugar), attention to glucose control is warranted during surgery as well as in the postoperative period. Consequently, measures to prevent and treat hyperglycemia - coupled with fasting status - places patients at considerable risk for perioperative hypoglycemia (low blood sugar). Outpatient patient studies support that profound hypoglycemia can be deleterious and even fatal to patients.

This descriptive study will utilize retrospective chart review to examine factors associated with hypoglycemia. Charts from 700 subjects who experienced blood glucose values less than 70 mg/dl primarily in the preoperative and postanesthesia care units at William Beaumont Hospital-Royal Oak will be reviewed. Another 1600 charts will be screened for subsequent intraoperative hypoglycemia: 800 that had low normal preoperative glucose values and 800 that had high preoperative values (with likelihood of insulin therapy).

Numerous factors believed to be associated with perioperative hypoglycemia will be analyzed including type and duration of diabetes, usual diabetes treatment regimen and alterations on day of surgery, self-reported usual fasting blood sugar range, duration of fasting, type of surgery and anesthesia, co-morbidities, and medications associated with hypoglycemia.

Determining factors associated with perioperative hypoglycemia will improve prediction of which patients are at highest risk for hypoglycemia, enabling healthcare providers to institute more conservative insulin therapy when indicated, initiate early maintenance intravenous dextrose, and/ or perform more frequent glucose testing. Identifying associated factors will improve hypoglycemic predictions and interventions which should lead to safer, more effective care for patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery at William Beaumont Hospital in Royal Oak, Michigan between January 1, 2003, and January 1, 2009.
* Point of care testing identified a blood sugar value less than 69 mg/dl at any time in the perioperative area; or a value between 70-89 mg/dl in the preoperative area; or a glucose value greater than 250 mg/dl in the preoperative area.

Exclusion Criteria:

* Obstetric patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon I Rosenblatt, MD, Principal Investigator — Michigan Endocrine Consultants; Tamra Dukatz, CRNA, Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective review of patients who underwent surgical procedures at our institution from 2003-2009
Pre-assignment Details: Retrospective
Groups:
- Low Normal Group: Patients with diabetes who arrived in preoperative area with blood glucose values of 70-89 mg/dl
- Hyperglycemia-treated Group: Patients with diabetes who had preoperative blood glucose values >249 mg/dl and were subsequently treated with insulin
Period: Overall Study
Arm/Group | Low Normal Group | Hyperglycemia-treated Group
Started | 308 (Retrospective review) | 279
Completed | 308 (Retrospective review) | 279
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Normal Group | Hyperglycemia-treated Group | Total
Number analyzed (Participants) | 308 | 279 | 587
Age Continuous [Mean (Standard Deviation); unit: years] | 61.34 (14.93) | 56.34 (14.18) | 58.96 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 137 | 279
  Male | 166 | 142 | 308
Region of Enrollment [Number; unit: participants]
  United States | 308 | 279 | 587
Diabetes type [Number; unit: participants]
  Type 1 diabetes | 37 | 47 | 84
  Type 2 diabetes | 217 | 175 | 392
  type not documented | 54 | 57 | 111
Renal disease [Number; unit: participants]
  Renal disease documented | 85 | 54 | 139
  Renal disease not documented | 223 | 225 | 448
Insulin regimen prior to preop arrival [Number; unit: participants]
  Insulin use | 266 | 240 | 506
  No documented insulin use | 42 | 39 | 81
Beta-blocker medication in regimen [Number; unit: participants]
  Documented Beta blocker use | 148 | 107 | 255
  No documented beta blocker use | 160 | 172 | 332

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Incidence
Description: Blood glucose values <70 mg/dl
Time Frame: perioperative period
Measure: Number; unit: participants
Arm/Group | Low Normal Group | Hyperglycemia-treated Group
Number analyzed (Participants) | 308 | 279
participants | 53 | 10
Statistical Analysis 1: Comparison: Low Normal Group vs Hyperglycemia-treated Group; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = .18, 95% CI 2-sided [.09 to .18], Standard Error of Mean .36

ADVERSE EVENTS:
Groups:
- Adverse Events Not Collected: Adverse Events Not Collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Point-of-care blood glucose testing was most often the means of measurement. Frequency of glucose monitoring was not standardized. Retrospective review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No